CLINICAL TRIAL: NCT05586737
Title: Effects of Immunomodulatory Therapy on Gonadal Function in Women With Autoimmune Premature Ovarian Insufficiency
Brief Title: Immunomodulatory Therapy in Women With Autoimmune Premature Ovarian Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Angelica Lindén Hirschberg (Other)
Responsible Party: Sponsor-Investigator, Angelica Lindén Hirschberg, Professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KarolinskaUniversityHospital
Record Dates: First submitted 2022-10-09; First posted 2022-10-19 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Autoimmune Diseases; Premature Ovarian Insufficiency
MeSH Terms: conditions — Autoimmune Diseases; Primary Ovarian Insufficiency | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- rituximab (Experimental): Controlled ovarian hyperstimulation will be performed before and four months after two infusions of 1-gram rituximab (Mabthera®).
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — 1 gram rituximab twice with two weeks interval

SUMMARY:
Title: Effects of immunomodulatory therapy on gonadal function in women with autoimmune premature ovarian insufficiency (POI)

Trial objectives and purpose: To study if rituximab therapy can improve ovarian response to gonadotropin stimulation and menstrual function in women with autoimmune POI.

Treatment: Controlled ovarian hyperstimulation before and four months after an infusion of 1-gram rituximab (Mabthera®) twice with two weeks interval. Follow-up period 12 months after infusion.

Primary outcome: Number of antral follicles and the size of the largest follicle in response to ovarian stimulation.

Secondary outcomes:

1. Reestablishment of spontaneous menstrual bleedings during the 12 months' study period
2. Ovulation during the 12 months' study period
3. Change in B-cell count, autoantibody indices and immunoglobulin levels (IgG) after treatment

Safety outcomes: All adverse events. Of particular relevance are any hospital admissions, infections and allergic reactions.

Study population: Fifteen women with autoimmune POI defined as absence of menstruation > 6 months and elevated serum level of follicle stimulation hormone > 40 International units (IU)/L.

Inclusion criteria: Autoimmune POI defined as presence of autoantibodies against 21-hydroxylase (OH), side chain cleavage enzyme (SCC), 17-OH and/or neuronal apoptosis inhibitory protein (NACHT) leucine-rich-repeat protein 5 (NALP5) or other relevant autoantibodies; 18-35 yrs of age; body mass index 19-30.

Exclusion criteria: Hypersensitivity to rituximab; severe infection; severe immunosuppression; cardiac disease; cancer; benign tumours of the hypothalamus, pituitary, or ovary; ovarian enlargement or ovarian cyst; vaginal bleeding of unknown aetiology.

Time plan: The study is expected to start the spring 2017. It is expected to be closed spring 2023.

ELIGIBILITY:
Inclusion Criteria:

1. Autoimmune premature ovarian insufficiency defined as presence of autoantibodies against 21-OH, SCC, 17-OH and/or NALP5 or other relevant autoantibodies
2. 18-35 yrs of age
3. Body mass index 19-30.
4. In fertile females, willingness to comply with effective contraceptive methods.
5. Ability to provide informed consent

Exclusion Criteria:

1. Documented hypersensitivity or intolerance to rituximab
2. Active, severe infection
3. Severe immunosuppression
4. Severe cardiac disease
5. Cancer
6. Benign tumours of the hypothalamus, pituitary, or ovary; ovarian enlargement or ovarian cyst
7. Vaginal bleeding of unknown aetiology
8. Hormone replacement therapy (HRT) within four weeks prior study entry.
9. Pregnant or lactating women
10. Concurrent treatment with other immunosuppressive drugs
11. Vaccination within 4 weeks of infusion of study medication
12. Severe psychiatric disorder
13. Patient with any condition or any circumstance that in the opinion of the investigator would make it unsafe to undergo treatment with Rituximab.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Number of antral follicles in response to ovarian stimulation 4 months after last rituximab infusion. | 4 months
  Vaginal ultrasound measurement
The largest follicle in response to ovarian stimulation 4 months after last rituximab infusion. | 4 months
  Vaginal ultrasound measurement

SECONDARY OUTCOMES:
Spontaneous menstrual bleedings during the 12 months' study period | 12 months
  Number of spontaneous menstrual bleedings
Ovulation during the 12 months' study period | 12 months
  Confirmed ovulation (y/n)
Immunoglobulin levels | 4 and 12 months
  Change in immunoglobulin levels (g/L) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Olle Kämpe, MD, PhD, Study Chair — Karolinska Institutet
Locations (1):
- Angelica Hirshberg, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No